CLINICAL TRIAL: NCT04530903
Title: Interest in Clonidine in Association With Levobupivacaine Performing a Pudendal Block in Proctological Surgery: Pilot Study, Prospective
Brief Title: Interest in Clonidine in Association With Levobupivacaine Performing a Pudendal Block in Proctological Surgery.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B076202042809
Record Dates: First submitted 2020-06-18; First posted 2020-08-28 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Proctological Surgery
Keywords: Post-operative Pain; Pudendal Block; Clonidine; Levobupivacaine
MeSH Terms: conditions — Pain, Postoperative | interventions — Clonidine; Levobupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Clonidine (Experimental): Group Clonidine will benefit from the pudendal block realised with 10 ml of 0.25% levobupivacaine and 75 µg of clonidine per side.
  Interventions: Drug: Clonidine; Drug: Levobupivacaine
- Control (Placebo Comparator): Group Control will benefit from the pudendal block realised with 10 ml of 0.25% levobupivacaine per side; 0.5 ml of 0.9% NaCl will be added to each syringe to homogenise the volume in order to remain blind.
  Interventions: Drug: Levobupivacaine; Drug: NaCl 0.9%

INTERVENTIONS:
Drug: Clonidine — 75 µg (0.5mL) per injection site
  Other Names: Catapressan
  Arms: Group Clonidine
Drug: Levobupivacaine — 0.25% (10 ml) per injection site
  Other Names: Chirocaine
Drug: NaCl 0.9% — Nacl 0.9% (0.5ml) per injection site
  Arms: Control

SUMMARY:
Proctological surgery represents a short duration surgery performed in ambulatory, which causes significant post-operative pain.

Post-operative pain resulting from proctological surgery is greater than 5 on the Visual Analog Scale (VAS) within the first 24 hours and it revives during the first defecation.

The ideal pain management procedures are based on the multimodal analgesia model, based in turn on the combination of products and / or techniques to improve the quality of analgesia, reduce the side effects linked to the use of opioids, reduce responses to surgical stress, reduce postoperative recovery and allow rapid rehabilitation of the patient.

The aim of our study is to investigate whether clonidine combined with levobupivacaine in the pudendal block reduce the total consumption of opioids in proctological surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signature of informed consent

Exclusion Criteria:

* Refusal to participate ;
* Allergy to either local anaesthetics or clonidine;
* Local infectious pathologies (e.g. acute ano-perineal suppuration)
* Pregnancy
* Breastfeeding
* Severe bradyarrhythmia due to sinus node disease or second and third degree atrioventricular block
* Severe depressive condition
* Severe coronary artery disease
* Raynaud's disease
* Heart failure
* Obliterating thromboangiitis
* Epilepsy
* Spinal anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Total Dose of Opioids consumed in the intraoperative period | up to 24 hours post-surgery
  Total consumption of sufentanyl during the intraoperative period (in micrograms). The administration of sufentanyl depends on the change of physiological parameters (augmentation of 20% of blood pressure and/or cardiac frequency).

SECONDARY OUTCOMES:
Total Dose of tramadol consumed in the recovery room | up to 24 hours post-surgery
  In the recovery room, dose of tramadol (in milligrams, intravenous administration). The administration of tramadol depends on Visual Analogic Pain Score (VAS>4) (scale = 0 no pain; 10 = worst pain imaginable)
Total consumption of tramadol in post-operative period | up to 24 hours post-surgery
  Total consumption of tramadol from the exit of the recovery room to the day after the surgery based on Visual Analogic Pain Score >4 (scale = 0 no pain; 10 = worst pain imaginable).
  Tramadol (dose in milligrams, oral administration)
Need for tramadol administration per patient during the first 24 hours | up to 24 hours post-surgery
  Number of Tramadol dose requested by the patient during the first 24 hours
Total Dose of piritramide consumed in the recovery room | up to 24 hours post-surgery
  In the recovery room, dose of piritramide (in milligrams, intravenous administration). The administration of piritramide depends on Visual Analogic Pain Score (VAS>4) (scale = 0 no pain; 10 = worst pain imaginable)
Need for Piritramid administration per patient during the hospitalization in Post Anesthesia Care Unit (PACU) | during the hospitalization in Post Anesthesia Care Unit (PACU)
  Number of Piritramid dose requested by the patient during the hospitalization in Post Anesthesia Care Unit (PACU)
Total consumption of paracetamol in post-operative period | up to 24 hours post-surgery
  Total consumption of paracetamol from the exit of the recovery room to the day after the surgery based on Visual Analogic Pain Score >4 (scale = 0 no pain; 10 = worst pain imaginable). Paracetamol (dose in grams, oral administration)
Total consumption of diclofenac in post-operative period | up to 24 hours post-surgery
  Total consumption of diclofenac from the exit of the recovery room to the day after the surgery based on Visual Analogic Pain Score >4 (scale = 0 no pain; 10 = worst pain imaginable).
  Diclofenac (dose in milligrams, oral administration)
Time before First Use of Rescue Analgesic | up to 24 hours post-surgery
  Time between the completion of the block and the first post-operative administration of rescue analgesics (Tramadol and/or Piritramide on request)
Post-operative Pain as assessed by Visual Analog Scale | up to 24 hours post-surgery
  Post-operative Pain levels will be determined every 15 minutes in the recovery room, then every hour until discharge and on Day 1 at home; Visual Analog pain score (scale = 0 no pain; 10= worst pain imaginable)
Patient satisfaction | up to 24 hours post-surgery
  Level of satisfaction assessed on a 5-point scale (from 1 to 5): 1 not satisfied, 2 not very satisfied, 3 moderately satisfied, 4 satisfied, 5 very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Panayota Kapessidou, MD,PhD, Study Director — University Hospital Saint-Pierre (CHU Saint-Pierre), Université Libre de Bruxelles (ULB); Myriam Suball, MD, Principal Investigator — University Hospital Saint-Pierre (CHU Saint-Pierre), Université Libre de Bruxelles (ULB); Marzia Gambassi, MD, Principal Investigator — University Hospital Saint-Pierre (CHU Saint-Pierre), Université Libre de Bruxelles (ULB)
Locations (1):
- University Hospital Saint-Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joshi GP. Multimodal analgesia techniques and postoperative rehabilitation. Anesthesiol Clin North Am. 2005 Mar;23(1):185-202. doi: 10.1016/j.atc.2004.11.010. PMID 15763418
- [Background] Ceulemans A, De Looze D, Van de Putte D, Stiers E, Coppens M. High post-operative pain scores despite multimodal analgesia in ambulatory anorectal surgery: a prospective cohort study. Acta Chir Belg. 2019 Aug;119(4):224-230. doi: 10.1080/00015458.2018.1500802. Epub 2018 Sep 7. PMID 30189793
- [Background] Joshi GP, Neugebauer EA; PROSPECT Collaboration. Evidence-based management of pain after haemorrhoidectomy surgery. Br J Surg. 2010 Aug;97(8):1155-68. doi: 10.1002/bjs.7161. PMID 20593430
- [Background] Comite douleur-anesthesie locoregionale et le comite des referentiels de la Sfar. [Formalized recommendations of experts 2008. Management of postoperative pain in adults and children]. Ann Fr Anesth Reanim. 2008 Dec;27(12):1035-41. doi: 10.1016/j.annfar.2008.10.002. Epub 2008 Nov 21. No abstract available. French. PMID 19026514
- [Background] Novikova N, Cluver C. Local anaesthetic nerve block for pain management in labour. Cochrane Database Syst Rev. 2012 Apr 18;2012(4):CD009200. doi: 10.1002/14651858.CD009200.pub2. PMID 22513972
- [Background] Vinson-Bonnet B.. Le bloc pudendal: technique d'analgésie postopératoire en chirurgie proctologique. Pelvi-Périnéologie 2007, 2(2):180-183.
- [Background] Naja Z, Ziade MF, Lonnqvist PA. Nerve stimulator guided pudendal nerve block decreases posthemorrhoidectomy pain. Can J Anaesth. 2005 Jan;52(1):62-8. doi: 10.1007/BF03018582. PMID 15625258
- [Background] Capdevila X, Barthelet Y, Biboulet P, Ryckwaert Y, Rubenovitch J, d'Athis F. Effects of perioperative analgesic technique on the surgical outcome and duration of rehabilitation after major knee surgery. Anesthesiology. 1999 Jul;91(1):8-15. doi: 10.1097/00000542-199907000-00006. PMID 10422923
- [Background] Imbelloni LE, Vieira EM, Gouveia MA, Netinho JG, Spirandelli LD, Cordeiro JA. Pudendal block with bupivacaine for postoperative pain relief. Dis Colon Rectum. 2007 Oct;50(10):1656-61. doi: 10.1007/s10350-007-0216-7. PMID 17701375
- [Background] De La Arena P.. Bloc pudendal sous échographie: faisabilité et efficacité peropératoire chez l'enfant. Annales Françaises d'Anesthésie et de Réanimation 2014; A398-A403.
- [Background] Gaudet-Ferrand I, De La Arena P, Bringuier S, Raux O, Hertz L, Kalfa N, Sola C, Dadure C. Ultrasound-guided pudendal nerve block in children: A new technique of ultrasound-guided transperineal approach. Paediatr Anaesth. 2018 Jan;28(1):53-58. doi: 10.1111/pan.13286. Epub 2017 Dec 5. PMID 29205687
- [Background] Li A, Wei Z, Liu Y, Shi J, Ding H, Tang H, Zheng P, Gao Y, Feng S. Ropivacaine versus levobupivacaine in peripheral nerve block: A PRISMA-compliant meta-analysis of randomized controlled trials. Medicine (Baltimore). 2017 Apr;96(14):e6551. doi: 10.1097/MD.0000000000006551. PMID 28383425
- [Background] Malav K, Singariya G, Mohammed S, Kamal M, Sangwan P, Paliwal B. Comparison of 0.5% Ropivacaine and 0.5% Levobupivacaine for Sciatic Nerve Block Using Labat Approach in Foot and Ankle Surgery. Turk J Anaesthesiol Reanim. 2018 Feb;46(1):15-20. doi: 10.5152/TJAR.2017.03411. Epub 2017 Nov 27. PMID 30140496
- [Background] Brummett CM, Williams BA. Additives to local anesthetics for peripheral nerve blockade. Int Anesthesiol Clin. 2011 Fall;49(4):104-16. doi: 10.1097/AIA.0b013e31820e4a49. PMID 21956081
- [Background] Kirksey MA, Haskins SC, Cheng J, Liu SS. Local Anesthetic Peripheral Nerve Block Adjuvants for Prolongation of Analgesia: A Systematic Qualitative Review. PLoS One. 2015 Sep 10;10(9):e0137312. doi: 10.1371/journal.pone.0137312. eCollection 2015. PMID 26355598
- [Background] Bernard JM, Macaire P. Dose-range effects of clonidine added to lidocaine for brachial plexus block. Anesthesiology. 1997 Aug;87(2):277-84. doi: 10.1097/00000542-199708000-00014. PMID 9286891
- [Background] Kelika P, Arun JM. Evaluation of clonidine as an adjuvant to brachial plexus block and its comparison with tramadol. J Anaesthesiol Clin Pharmacol. 2017 Apr-Jun;33(2):197-202. doi: 10.4103/joacp.JOACP_58_13. PMID 28781445
- [Background] Popping DM, Elia N, Marret E, Wenk M, Tramer MR. Clonidine as an adjuvant to local anesthetics for peripheral nerve and plexus blocks: a meta-analysis of randomized trials. Anesthesiology. 2009 Aug;111(2):406-15. doi: 10.1097/ALN.0b013e3181aae897. PMID 19602964
- [Background] McCartney CJ, Duggan E, Apatu E. Should we add clonidine to local anesthetic for peripheral nerve blockade? A qualitative systematic review of the literature. Reg Anesth Pain Med. 2007 Jul-Aug;32(4):330-8. doi: 10.1016/j.rapm.2007.02.010. PMID 17720118